CLINICAL TRIAL: NCT05987059
Title: Involving Communities in Addressing the Maternal Health Crisis: Making an IMPACT
Acronym: Project IMPACT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Morehouse School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: MH-CIP Project IMPACT
Record Dates: First submitted 2023-06-30; First posted 2023-08-14 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2024-11

CONDITIONS: Preconception Health

STUDY DESIGN:
Intervention Model Description: The proposed study will be a Type 2 hybrid effectiveness-implementation RCT with individual level randomization to one of two intervention study arms (standard and enhanced implementation strategy packages) in years 2-4 and data from a non-randomized third study arm (control group) captured in year 1. An expected 10 community-based organizations will participate in the study. A hybrid type 2 design is ideal because there are effectiveness studies conducted on preconception counseling conducted in clinical settings, but there is still a dearth of evidence on both effectiveness and implementation of preconception counseling in community-based settings and specifically with Black women and in Black-led organizations. The hybrid type 2 design would allow for continued evaluation of the effectiveness of the intervention and could capitalize on the implementation occurring to evaluate the impact of implementation strategies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Structured Follow-Up (Experimental): Emailed informational flyer(s) on prioritized cardiovascular risks and text messaging for logistical reasons. These will be in addition to the SBIRT intervention delivered by Healthy Start and other similar community organization staff that all participants will receive.
  Interventions: Behavioral: SBIRT Intervention
- Enhanced Structured Follow-Up (Experimental): Text or phone message(s) focused on the same prioritized risks + emailed informational flyer(s). These will be in addition to the SBIRT intervention delivered by Healthy Start and other similar community organization staff that all participants will receive.
  Interventions: Behavioral: SBIRT Intervention

INTERVENTIONS:
Behavioral: SBIRT Intervention — Project IMPACT intervention will follow a Screening, Brief Intervention, and Referral to Treatment (SBIRT) Model. In the proposed study, staff at community sites will deliver a tailored SBIRT model for people seeking to get pregnant as our "Project IMPACT intervention". SBIRT was originally developed as a public health model designed to provide universal screening, secondary prevention (detecting risky or hazardous substance use before the onset of abuse or dependence), early intervention, and treatment for people who have problematic or hazardous alcohol problems within primary care and other health care settings. Morehouse School of Medicine (MSM) has adapted this SBIRT model for people who are seeking to get pregnant to assess their risks and provide early intervention to at-risk people of reproductive age who want to get pregnant. Brief preconception counseling interventions addressing multiple behavioral risk factors have been found to be effective in prior studies.

SUMMARY:
With support from the National Heart, Lung, and Blood Institute, The Center for Maternal Health Equity at Morehouse School of Medicine is conducting a research study to test the implementation of Pre-Pregnancy Counseling in community-based settings.

DETAILED DESCRIPTION:
Severe racial disparities in pregnancy-related cardiovascular morbidity and mortality are preventable and warrant timely community-engaged action. Black women are 3 times more likely to die from a pregnancy-related cause, as compared to white women10 -in part, due to higher rates of cardiovascular risk during pregnancy. More than 80% of pregnancy-related deaths in the U.S. are preventable. Preconception counseling has been shown to improve maternal health for all women, with clear benefits to address cardiovascular risk factors of obesity, diabetes, hypertension. In order to have impact, evidence-based preconception counseling programs must be delivered through community settings that have a mission to reach at-risk populations of women. Healthy Start/community-based settings are appropriate for this, as they serve an at-risk population of Black women in many locations nationally. The investigators have engaged with Healthy Start and similar community-based settings in Georgia, South Carolina, to identify preconception counseling interventions that are evidence-based and feasible for their staff and community members. This community-engaged approach identified Screening, Brief Intervention, and Referral to Treatment (SBIRT) interventions as feasible and acceptable to both staff and patients. In the pilot-test of their SBIRT model approach (Project IMPACT intervention), the investigators demonstrated capacity to screen for pregnancy risks and provide early intervention to n = 23 at-risk persons of reproductive age who wanted to get pregnant within the year. The investigators will build on their pilot work to conduct a hybrid effectiveness/implementation trial (type 2 hybrid) with n = 10 sites serving low-income African American men and women in Georgia, NC, SC, and TN. The investigators will use EPIS as an overarching framework to guide progress across the four phases (exploration, preparation, implementation and sustainment). In Aim 1 (EPIS Preparation phase), the investigators will work with their community partners to tailor the implementation strategy packages (Aim 1a) and their Project IMPACT intervention (Aim 1b) to the context of 10 sites across 4 states -- this tailoring will address contextual determinants of successful implementation from the Pragmatic Robust Implementation and Sustainability Model (PRISM). In Aim 2 (EPIS Implementation phase), we will test an Enhanced vs. Standard implementation strategy package of structured follow-up on the number of pre-conception counseling visits completed and will test any structured follow-up vs. no structured follow-up on readiness to change for key cardiovascular risk factors. In Aim 3 (EPIS Sustainment phase), the investigators will work with their community sites to co-develop an implementation and sustainment guide for the most effective strategy bundle from Aim 2. This work has potential to impact racial disparities in pregnancy-related morbidity/mortality and to advance our collective scientific understanding of the relative benefits of alternate implementation strategy packages.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Black/ African-American
* Fluent English-Speaker
* Not pregnant at the time of enrollment
* Own a phone
* Receive services at the community-based site

Exclusion Criteria:

-

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 850 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Implementation | 6 months
  Each participant will remain in the study for six months and will complete three interviews (baseline, 3-month, 6-month follow-up). The number of pre-conception counseling sessions received by community members in the standard and enhanced intervention arms will be captured at 6 months. The proposed range for the primary implementation outcome will be 0-7 visits/contacts.
Effectiveness | baseline, 3 months, 6 months
  1) 0-10 readiness ruler (inclusive of all 5 stages of change)
  Each participant will remain in the study for six months and will complete three interviews (baseline, 3-month, 6-month follow-up). The stage of change score will be captured at baseline, 3 and 6 months. A text message reminder will be sent to patients at 3 and 6 months to help minimize missing data. The stage of change score will be captured for control subjects in year 1 and intervention subjects during the implementation phase. All participants from both implementation strategies will be combined into one group, and this group will be compared to the control group participants.
Effectiveness | baseline, 3 months, 6 months
  2) 0-10 readiness ruler (inclusive of all 5 stages of change)
  Each participant will remain in the study for six months and will complete three interviews (baseline, 3-month, 6-month follow-up). The stage of change score will be captured at baseline, 3 and 6 months. A text message reminder will be sent to patients at 3 and 6 months to help minimize missing data. The stage of change score will be captured for control subjects in year 1 and intervention subjects during the implementation phase. All participants from both implementation strategies will be combined into one group, and this group will be compared to the control group participants.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie D. Hernandez, PhD, Principal Investigator — Associate Professor; Cheryl Franklin, MD, Principal Investigator — AssociateProfessor; Oluyemi Farinu, PhD, Study Director — Project Director
Locations (1):
- Morehouse School of Medicine, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costanza-Chock S. Design justice: Community-led practices to build the worlds we need. The MIT Press; 2020.
- [Background] Wallerstein N, Duran B, Oetzel JG, Minkler M. On community-based participatory research. Community-based participatory research for health: Advancing social and health equity. 2017;3:3-16.
- [Background] Aguilar-Gaxiola S, Ahmed SM, Anise A, Azzahir A, Baker KE, Cupito A, Eder M, Everette TD, Erwin K, Felzien M, Freeman E, Gibbs D, Greene-Moton E, Hernandez-Cancio S, Hwang A, Jones F, Jones G, Jones M, Khodyakov D, Michener JL, Milstein B, Oto-Kent DS, Orban M, Pusch B, Shah M, Shaw M, Tarrant J, Wallerstein N, Westfall JM, Williams A, Zaldivar R. Assessing Meaningful Community Engagement: A Conceptual Model to Advance Health Equity through Transformed Systems for Health: Organizing Committee for Assessing Meaningful Community Engagement in Health & Health Care Programs & Policies. NAM Perspect. 2022 Feb 14;2022:10.31478/202202c. doi: 10.31478/202202c. eCollection 2022. No abstract available. PMID 35891775
- [Background] Surgo Ventures - The US Maternal Vulnerability Index (MVI). mvi.surgoventures.org. Published 2021. Accessed February 2023. https://mvi.surgoventures.org/
- [Background] Armstrong-Mensah E, Dada D, Bowers A, Muhammad A, Nnoli C. Geographic, Health Care Access, Racial Discrimination, and Socioeconomic Determinants of Maternal Mortality in Georgia, United States. Int J MCH AIDS. 2021;10(2):278-286. doi: 10.21106/ijma.524. Epub 2021 Dec 13. PMID 34938596
- [Background] Maternal, Child, and Infant Health. Mecknc.gov. Published 2019. Accessed February 4, 2023. https://www.mecknc.gov/HealthDepartment/HealthStatistics/Pages/MaternalChildInfantHealth.aspx